CLINICAL TRIAL: NCT04065321
Title: Effect of Circulating Tumor Cell Detection in Patients With Luminal A Breast Cancer Without Lymph Node Metastasis Instead of Conventional Imaging Examination After Operation: a Non-Inferiority Randomized Controlled Clinical Trial
Brief Title: Circulating Tumor Cell Detection in Patients With Luminal A Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Jianyi Li, Principal Investigator, Shengjing Hospital
Other Study IDs: Shengjing-LJY04
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Breast Neoplasms
Keywords: Circulating tumor cells; PET
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 250 patients will be assigned into control group.
  Interventions: Procedure: PET-CT examination
- Trial group: 250 patients will be assigned into trial group.
  Interventions: Procedure: Peripheral blood detection

INTERVENTIONS:
Procedure: PET-CT examination — All patients in the control group will undergo PET-CT examination after operation, and will reexamination once every 4 months in 2 years, every 6 months in 3-5 years, and every year in more than 5 years.
  Groups: Control group
Procedure: Peripheral blood detection — All patients in the trial group will be followed up after operation, and will reexamination once every 4 months in 2 years, every 6 months in 3-5 years, and every year in more than 5 years. Peripheral blood will be collected for detection of circulating tumor cells at each follow-up. If circulating tumor cells are abnormal (number of circulating tumor cells ≥ 2 or CD133 ≥ 1), PET-CT will be performed immediately.
  Groups: Trial group

SUMMARY:
The incidence of breast cancer in Chinese women has increased year by year, and luminal A breast cancer commonly occurs in early-stage and postmenopausal women. This type of breast cancer is not sensitive to chemotherapy, although it has a low mortality rate and distant metastasis rate. Studies have shown that luminal A breast cancer is sensitive to endocrine therapy. Patients with breast cancer who undergo excision should be followed up and their prognosis should be monitored regularly. At present, imaging detection is mainly used in the conventional follow-up of breast cancer, but the cost of many imaging examinations is high, so a cost-effective examination is urgently needed.

Recent studies have found that circulating tumor cells can be used as a new type of tumor molecular marker, which can be used to diagnose tumors, judge the prognosis and monitor the efficacy by detecting the number and characteristic protein expression of circulating tumor cells. Because circulating tumor cells may develop abnormalities 4-6 months earlier than conventional imaging examination, as long as circulating tumor cells of patients are abnormal, timely PET-CT examination will neither miss diagnosis nor delay the condition. Simultaneously, the cost of hospitalization can be obviously reduced.

This non-inferiority randomized controlled clinical trial is designed to compare the differences in postoperative conditions between circulating tumor cell detection and conventional imaging examination in patients with luminal A breast cancer without lymph node metastasis.

DETAILED DESCRIPTION:
Breast cancer ranks first in the incidence of female malignant tumors and second in mortality. It is mainly classified into luminal A, luminal B, human epidermal growth factor receptor 2 positive, basal-like and other special types of breast cancer. Epidemiological studies have shown that the incidence of luminal A breast cancer is 44.5-69.0%, mostly in early-stage patients and postmenopausal women, with a low mortality rate and distant metastasis rate. Luminal A breast cancer is usually invasive. Although it is not sensitive to chemotherapy, luminal A breast cancer is sensitive to endocrine therapy. Therefore, the treatment of luminal A breast cancer is a combination of surgery, chemotherapy, radiotherapy and endocrine therapy.

After surgical removal of breast cancer, follow-up should be conducted according to the National Comprehensive Cancer Network guidelines to monitor the prognosis at any time. Conventional follow-up is mainly based on imaging examination, but the cost of many imaging examinations is high, so a cost-effective examination is urgently needed.

Circulating tumor cells are tumor cells that fall off from solid tumors (primary and metastatic foci) and enter the peripheral blood. In recent 30 years, circulating tumor cells have become one of the new tumor molecular markers. Detection of the number and protein expression of circulating tumor cells can diagnose the disease, judge the prognosis and monitor the therapeutic effect. Epithelial-mesenchymal transition and overexpression of epithelial cell adhesion molecule in circulating tumor cells suggest that the prognosis of cancer patients is not good. By comparing the number of circulating tumor cells in blood before and after surgery or radiotherapy and chemotherapy,whether the treatment is effective or not can be judged, which has important clinical research and application value. Currently, many clinical trials have used circulating tumor cells to monitor the prognosis in breast cancer. Circulating tumor cells may develop abnormalities 4-6 months earlier than conventional imaging examination, and PET-CT can only find subclinical lesions 4-6 weeks in advance. Thus, as long as circulating tumor cells of patients are abnormal, timely PET-CT examination will neither miss diagnosis nor delay the condition. Simultaneously, the cost of hospitalization can be obviously reduced.

This non-inferiority randomized controlled clinical trial is designed to compare the differences in postoperative conditions between circulating tumor cell detection and conventional imaging examination in patients with luminal A breast cancer without lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

* estrogen receptor (≥ 10%), progesterone receptor (≥ 10%) and epidermal growth factor receptor 2 negative;
* proliferation index Ki-67 < 20%;
* no lymph node metastasis;
* systemic therapy (chemotherapy, radiotherapy and endocrine therapy) in accordance with the National Comprehensive Cancer Network guidelines;
* provision of informed consent of patients and their families.

Exclusion Criteria:

* Bilateral breast cancer;
* inflammatory breast cancer;
* pregnancy or lactation;
* history of other cancers or chest radiotherapy.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: 500 patients will be recruited from outpatients and admission office of Shengjing Hospital of China Medical University by posting recruitment notice listing the study details on the bulletin board. The patients will be randomly divided into trial group and control group, with 250 patients per group.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival refers to the period from breast cancer excision to local recurrence, distant metastasis confirmed by clinical evidence, diagnosis of the second primary tumor or death of the patient.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival refers to the time from breast cancer excision to death due to any cause

OTHER OUTCOMES:
Total length of hospital stay | 5 years
  Total length of hospital stay for patients during the reexamination
Average length of hospital stay per reexamination | 5 years
  Average length of hospital stay per reexamination = total length of hospital stay/number of reexaminations
Total cost of reexaminations | 5 years
  Total cost of all reexaminations, including medical insurance and other insurance reimbursements
Average cost per reexamination | 5 years
  Average cost per reexamination = total cost of reexaminations/number of reexaminations

CONTACTS AND LOCATIONS:
Overall Officials: Jianyi Li, MD, Principal Investigator — Shengjing Hospital
Locations (2):
- China (2):
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Cancer Hospital of China Medical University, Liaoning Cancer Hospital and Institute, Shenyang, Liaoning